CLINICAL TRIAL: NCT01281917
Title: A Phase II Study of Velcade and Temsirolimus for Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Study of Velcade and Temsirolimus for Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO10407; H-2010-0393 (Other: IRB); NCI-2011-00647 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2017-07

CONDITIONS: Non-Hodgkins Lymphoma
Keywords: velcade; temsirolimus; non-hodgkins lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bortezomib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade plus Temsirolimus (Experimental): Velcade 1.6 mg/m2 weekly (days 1, 8, 15, and 22) Temsirolimus 25mg IV weekly (days 1, 8, 15, 22, and 29)
  Treat for up to 6 cycles, cycles are 35 days long.
  Interventions: Drug: Velcade; Drug: Temsirolimus

INTERVENTIONS:
Drug: Velcade — Velcade, 1.6 mg/m2 weekly (days 1, 8, 15, and 22)
  Other Names: bortezomib, PS-341
Drug: Temsirolimus — Temsirolimus 25mg IV weekly (days 1, 8, 15, 22, and 29)
  Other Names: Torisel

SUMMARY:
The investigators want to find out if the drugs Velcade and temsirolimus given together are effective in treating cancer. Velcade and temsirolimus are each FDA approved individually for certain types of cancer (Velcade for multiple myeloma and mantle cell lymphoma, and temsirolimus for renal cell carcinoma) but are not currently approved in combination for B-cell non-Hodgkin lymphoma. The investigators are trying to find out if giving these 2 drugs together will improve the period of time that the patient's cancer is stopped or slowed from growing and causing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-cell non-Hodgkin lymphoma which includes: diffuse large B-cell lymphoma; primary mediastinal large B-cell lymphoma; follicular lymphoma (grade 1, 2 or 3); mantle cell lymphoma; small lymphocytic lymphoma; marginal zone lymphoma; lymphoplasmacytic lymphoma; B-cell lymphoblastic lymphoma; or Burkitt lymphoma. "Grey-zone" lymphomas must be approved by the Wisconsin Oncology Network (WON) Study Chair or Principal Investigator prior to enrollment.
* At least one measurable tumor mass (>1.5 cm in the long axis and > 1.0 cm in the short axis) that has not been previously irradiated, or has grown since previous irradiation.
* Documented relapse or progression following prior antineoplastic therapy.
* No clinical or documented radiographic evidence of central nervous system lymphoma.
* Eastern Cooperative Oncology Group [ECOG] performance status of 0-2.
* The following clinical laboratory values within 14 days prior to enrollment:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109 cells / L
* Platelets ≥ 100 x 109 cells / L
* Alanine transaminase (ALT) and Aspartate transaminase (AST) ≤ 3X the upper limit of normal (ULN)
* Total bilirubin ≤ 2X the upper limit of normal (ULN).
* Calculated creatinine clearance ≥40 mL/min (using the Cockcroft-Gault equation).
* Female subjects must be either post-menopausal for at least 1 year or surgically sterilized, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of Velcade, or agree to completely abstain from heterosexual intercourse.
* Male subjects, even if surgically sterilized (ie, status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusions:

* Antineoplastic, experimental, or radiation therapy within 14 days prior to enrollment, or 21 days prior to Day 1 of Cycle 1.
* Radioimmunoconjugates within 10 weeks of Day 1 of Cycle 1.
* Autologous stem cell transplant within 3 months before Day 1 of Cycle 1, or any prior history of allogeneic stem cell transplant.
* Platelet transfusion within 7 days of Day 1 of Cycle 1.
* Ongoing therapy with glucocorticoids. Prednisone ≤15 mg per day or its equivalent is allowed.
* Patient has Grade 2 or greater peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient has hypersensitivity to Velcade, boron or mannitol.
* Female subjects that are pregnant or breast-feeding.
* Serious medical or psychiatric illness that is likely to interfere with participation
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Prior therapy with both Velcade and temsirolimus. Patients who have previously been treated with either Velcade or temsirolimus (but not both) are eligible.
* Radiation therapy within 3 weeks before randomization.
* Patients must not be taking the following strong CyP3A inducers at study entry: phenytoin, phenobarbital, rifampin, carbamazepin, rifabutin, rifampicin, a one week washout period is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad S Kahl, MD, Principal Investigator — Universtity of Wisconsin- Madison; Timothy S Fenske, MD, Study Chair — Medical College of Wisconsin
Locations (18):
- United States (18):
  - Rapid City Regional Hospital John T. Vucurevich Cancer Care Institute, Rapid City, South Dakota
  - Aurora Baycare Medical Center-GreenBay, Green Bay, Wisconsin
  - St Vincent Regional Cancer Center CCOP, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Inc, Green Bay, Wisconsin
  - Gunderson Lutheran Health System, La Crosse, Wisconsin
  - UW Health Oncology- 1 S Park, Madison, Wisconsin
  - University Of Wisconsin Cancer Center, Madison, Wisconsin
  - Aurora BayCare Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Columbia St Mary's, Inc, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sheboygan Memorial Medical Center, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aurora Medical Center in Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin
  - Aurora Health Care Metro, Inc., Wauwatosa, Wisconsin
  - UW Cancer Center-Riverview, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with relapsed or refractory B-cell NHL were enrolled from 10 sites within the Wisconsin Oncology Network (WON) between May 2011 and May 2013.
Pre-assignment Details: Forty participants were enrolled from 10 sites within the Wisconsin Oncology Network (WON) over 2 years. One participant withdrew consent immediately after enrollment and was never treated. Therefore, results are reported on the remaining 39 participants.
Groups:
- Velcade Plus Temsirolimus: Velcade 1.6 mg/m2 weekly (days 1, 8, 15, and 22) Temsirolimus 25mg IV weekly (days 1, 8, 15, 22, and 29)
  Treat for up to 6 cycles, cycles are 35 days long.
  Velcade: Velcade, 1.6 mg/m2 weekly (days 1, 8, 15, and 22)
  Temsirolimus: Temsirolimus 25mg IV weekly (days 1, 8, 15, 22, and 29)
Period: Overall Study
Arm/Group | Velcade Plus Temsirolimus
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The study enrolled patients with relapsed and refractory B-cell non-Hodgkin lymphoma.
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 68 [38 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 39
Number of prior treatments [Median (Full Range); unit: Prior treatments] | 4 [1 to 11]
Histology [Count of Participants; unit: Participants]
  DLBCL | 18
  Follicular lymphoma | 9
  Mantle cell lymphoma | 7
  Small lymphocytic lymphoma | 3
  Marginal zone lymphoma | 2
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG scales and criteria are used by doctors and researchers to assess how a patient's disease is progressing. Grade 0 is no affect to the daily living abilities of the patient, and Grade 5 is dead. This study was limited to participants with ECOG grades 0-2. Grade 0 is "Fully active, able to carry on all pre-disease performance without restriction," and Grade 2 is "Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours."
  Participants
    0 | 17
    1 | 16
    2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The primary objective of this study is to determine whether Velcade in combination with temsirolimus provides benefit to subjects with relapsed or refractory B-cell non-Hodgkin lymphoma as assessed by overall response rate (ORR) to therapy. ORR is the sum of patients with a Complete Response and Partial Response to therapy. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete REsponse (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 60 months
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
Percentage of participants | 31 [17 to 46.6]

2. Primary Outcome: Progression Free Survival
Description: The primary objective of this study is to determine whether Velcade in combination with temsirolimus provides benefit to subjects with relapsed or refractory B-cell non-Hodgkin lymphoma as assessed by progression-free survival (PFS).
Time Frame: Up to 60 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
Months | 4.7 [2.9 to 7.8]

3. Secondary Outcome: Safety of This Regimen
Description: Safety of the regimen will be measured by frequency and severity of adverse events.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
Participants
  Grade 3 Adverse Events | 31
  Grade 4 Adverse Events | 2
  No Grade 3/4 Adverse Events | 6

4. Secondary Outcome: Complete Response Rate
Description: The complete response rate (CR) to therapy as defined by International Lymphoma Response Criteria.
Time Frame: Up to 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
Participants | 3

5. Secondary Outcome: Tolerability of the Regimen
Description: Tolerability of the regimen is measured by the number of subjects able to complete the therapy as planned.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
Participants
  Discontinued study due to an adverse event | 5
  Continued study | 34

6. Secondary Outcome: Duration of Response
Description: Duration of Response is how long a response to therapy is held before a subject has progressive disease.
Time Frame: Up to 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
months | 7 [5.2 to 999]

7. Secondary Outcome: Overall Survival
Description: Length of time from enrollment until death.
Time Frame: Up to 60 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade Plus Temsirolimus
Number analyzed (Participants) | 39
Months | 14.1 [5.0 to 999]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 3 years and 1 month.
Description: Adverse events were graded at each evaluation and are reported according to version 4 of the National Cancer Institute's Common Terminology Criteria for Adverse Events.
Arm/Group | Velcade Plus Temsirolimus
All-Cause Mortality (participants affected / at risk) | 16/39
Serious Adverse Events (participants affected / at risk) | 18/39
Other Adverse Events (participants affected / at risk) | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade Plus Temsirolimus (N=39)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Heart Failure (Cardiac disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Palsy (right side of face) (Nervous system disorders) | 1 (1)
Scrotal Pain (Reproductive system and breast disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Shaking chills/non neutropenic fever and chills (Blood and lymphatic system disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Temsirolimus (Blood and lymphatic system disorders) | 1 (1)
Thrombolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade Plus Temsirolimus (N=39)
Platelet count decreased (Investigations) | 24 (82)
Fatigue (General disorders) | 20 (36)
Neutrophil count decreased (Investigations) | 18 (46)
Nausea (Gastrointestinal disorders) | 18 (27)
Diarrhea (Gastrointestinal disorders) | 17 (32)
Anorexia (Metabolism and nutrition disorders) | 16 (22)
Anemia (Blood and lymphatic system disorders) | 13 (29)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Vomiting (Gastrointestinal disorders) | 11 (15)
Chills (General disorders) | 11 (20)
Edema limbs (General disorders) | 11 (18)
White blood cell decreased (Investigations) | 10 (28)
Constipation (Gastrointestinal disorders) | 10 (12)
Dizziness (Nervous system disorders) | 10 (13)
Mucositis oral (Gastrointestinal disorders) | 9 (12)
Lymphocyte count decreased (Investigations) | 8 (19)
Abdominal pain (Gastrointestinal disorders) | 8 (11)
Headache (Nervous system disorders) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (9)
Insomnia (Psychiatric disorders) | 8 (10)
Fever (General disorders) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Infections and infestations - Other (Infections and infestations) | 6 (7)
Hypotension (Vascular disorders) | 6 (7)
Dysgeusia (Nervous system disorders) | 5 (5)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6)
Hypokalemia (Metabolism and nutrition disorders) | 4 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Creatinine increased (Investigations) | 3 (3)
Investigations - Other, specify (Investigations) | 3 (9)
Weight loss (Investigations) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
Ataxia (Nervous system disorders) | 3 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (4)
Paresthesia (Nervous system disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Lung infection (Infections and infestations) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 3 (3)
Blurred vision (Eye disorders) | 3 (4)
Conjunctivitis (Eye disorders) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Cholesterol high (Investigations) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 2 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 2 (2)
Peripheral nerve infection (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 2 (4)
Heart failure (Cardiac disorders) | 2 (2)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes